CLINICAL TRIAL: NCT03120637
Title: Evaluating in Cirrhotics With Refractory Vasoplegia the Effect of Methylene Blue in Sepsis: A Randomized Controlled Trial
Brief Title: Evaluating in Cirrhotics With Refractory Vasoplegia the Effect of Methylene Blue
Acronym: CRuMBS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: ILBS-Septic Shock-01
Record Dates: First submitted 2017-02-28; First posted 2017-04-19 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Septic Shock; Vasoplegia; Cirrhosis, Liver; Refractory Shock
Keywords: Methylene Blue; Septic Shock; Vasoplegia; Cirrhosis
MeSH Terms: conditions — Shock, Septic; Vasoplegia; Liver Cirrhosis; Shock; Fibrosis | interventions — Methylene Blue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylene Blue (Experimental): Methylene Blue intravenous route, 2 mg/kg Loading Dose over 30 minutes, followed by 0.5 mg/kg/hr for 6 hours
  Interventions: Drug: Methylene Blue
- Standard Treatment (No Intervention)

INTERVENTIONS:
Drug: Methylene Blue
  Arms: Methylene Blue

SUMMARY:
Mortality rates associated septic shock remains unacceptably high, around 20-50%, with refractory hypotension in half of these patients. Widespread vasodilatation involves the activation of the soluble intracellular enzyme guanylate cyclase (GC) by nitric oxide (NO), resulting in the production of cyclic guanosine monophosphate (cGMP). Initially discovered as an endothelium-derived relaxing factor in blood vessels, NO is made by the enzyme nitric oxide synthase (NOS). It has been suggested that the inhibition of NO generation might be a treatment option for sepsis and septic shock. Methylene blue (MB) is a dye that easily crosses cell membranes, inhibits iNOS, and is capable of inhibiting the GC enzyme in vascular smooth muscle cells.Early use of MB can block the progressive decrease in systemic vascular resistance of patients unresponsive to noradrenaline and mitigate the need for prolonged vasoconstrictor use. The investigators propose to study the effect of methylene blue on cirrhotic adults with sepsis, with refractory vasoplegia unresponsive to maximum doses of noradrenaline and vasopressin.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 years )
2. Refractory septic shock (Noradrenaline >0.5mcg/kg/mt )

Exclusion Criteria:

1. Declined consent
2. Pregnancy
3. Less than 18 years old
4. Immunosuppressant patients (e.g. on steroid medication, active anti-cancer chemotherapeutic agent, etc.)
5. Glucose-6-phosphate dehydrogenase deficiency
6. Medication of Serotonin modulator/SSRI
7. Pre-existing Pulmonary Hypertension
8. CKD-Stage IV/V
9. Patients with GI bleed
10. Patients on DNR
11. Patients declared Brain dead

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Survival in both groups | 2 days

SECONDARY OUTCOMES:
Systemic Vascular Resistance | 6 hours
  Change in SVR
Mean Arterial Pressure | 6 hours
  Improvement in MAP
Decrease of vasopressor dose of 20 percent from time of start of test drug. | 6 hours
  Effect on decreasing vasopressor doses

CONTACTS AND LOCATIONS:
Overall Officials: Karthik Ponnappan, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Liver Coma ICU, Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bassi E, Park M, Azevedo LC. Therapeutic strategies for high-dose vasopressor-dependent shock. Crit Care Res Pract. 2013;2013:654708. doi: 10.1155/2013/654708. Epub 2013 Sep 15. PMID 24151551
- [Result] Park BK, Shim TS, Lim CM, Lee SD, Kim WS, Kim DS, Kim WD, Koh Y. The effects of methylene blue on hemodynamic parameters and cytokine levels in refractory septic shock. Korean J Intern Med. 2005 Jun;20(2):123-8. doi: 10.3904/kjim.2005.20.2.123. PMID 16134766
- [Result] Kirov MY, Evgenov OV, Evgenov NV, Egorina EM, Sovershaev MA, Sveinbjornsson B, Nedashkovsky EV, Bjertnaes LJ. Infusion of methylene blue in human septic shock: a pilot, randomized, controlled study. Crit Care Med. 2001 Oct;29(10):1860-7. doi: 10.1097/00003246-200110000-00002. PMID 11588440
- [Result] Memis D, Karamanlioglu B, Yuksel M, Gemlik I, Pamukcu Z. The influence of methylene blue infusion on cytokine levels during severe sepsis. Anaesth Intensive Care. 2002 Dec;30(6):755-62. doi: 10.1177/0310057X0203000606. PMID 12500513
- [Result] Juffermans NP, Vervloet MG, Daemen-Gubbels CR, Binnekade JM, de Jong M, Groeneveld AB. A dose-finding study of methylene blue to inhibit nitric oxide actions in the hemodynamics of human septic shock. Nitric Oxide. 2010 May 15;22(4):275-80. doi: 10.1016/j.niox.2010.01.006. Epub 2010 Jan 28. PMID 20109575